CLINICAL TRIAL: NCT03045276
Title: Urological and Renal Disease Engaging Adolescents in Adherence Collaborative Trial
Acronym: U-REAACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Boston Children's Hospital (Other); Children's Healthcare of Atlanta (Other); Children's Mercy Hospital Kansas City (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-013000; 1R01DK110749 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Spina Bifida; Kidney Transplant
Keywords: Spina Bifida; Kidney Transplant
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - No Feedback, Minimum Incentive (Active Comparator): Subjects will receive daily text message reminders and report real-time treatment adherence with photos. They will receive compensation to encourage real-time adherence reporting. Subjects will also be able to log into a personal dashboard with a visual display of their weekly adherence performance and educational resources related to their primary disease. Every month, participants will receive a text encouraging them to visit their personal dashboard. The dashboard is able to track usage of the modules by individual. Parents/legal guardians will have access to these same educational materials via their own portals. Additionally, to mitigate the minimal risk of this study, parents/legal guardians will be notified if their child is excessively non-adherent.
  Interventions: Behavioral: Behavioral Feedback and Economic Incentives: Arm 1
- Arm 2 - Feedback, Maximum Incentive (Active Comparator): Subjects will receive daily text message reminders and report real-time treatment adherence with photos, and will have web access to the educational modules through their portal. Every month, participants will receive a text encouraging them to visit their portals. In contrast to Arm 1, they will receive their weekly performance results by text to their phone with tailored feedback. In Arm 2, subjects will receive a larger incentive if they perform their desired treatment behavior. Incentive notification will be texted to participants. Similarly to Arm 1, parents/legal guardians will have access to the same educational materials via their own WTH portals. Additionally, to mitigate the minimal risk of this study, parents/legal guardians will be notified if their child is excessively non-adherent.
  Interventions: Behavioral: Behavioral Feedback and Economic Incentives: Arm 2

INTERVENTIONS:
Behavioral: Behavioral Feedback and Economic Incentives: Arm 1 — The purpose of this study is to determine the effectiveness of behavioral feedback plus economic incentives to promote treatment adherence among a large diverse population of adolescents and young adults (AYA) with kidney transplants (KT) or spina bifida (SB). In Arm 1, participants will not receive personalized feedback, nor will they receive the "extra" incentive of $10 for meeting their adherence goal.
  Arms: Arm 1 - No Feedback, Minimum Incentive
Behavioral: Behavioral Feedback and Economic Incentives: Arm 2 — The purpose of this study is to determine the effectiveness of behavioral feedback plus economic incentives to promote treatment adherence among a large diverse population of adolescents and young adults (AYA) with kidney transplants (KT) or spina bifida (SB). In Arm 2, participants will receive personalized feedback, and an "extra" incentive of $10 for meeting their adherence goal.
  Arms: Arm 2 - Feedback, Maximum Incentive

SUMMARY:
The purpose of this study is to determine the effectiveness of behavioral feedback plus economic incentives to promote treatment adherence among a large diverse population of adolescents and young adults (AYA) with kidney transplant (KT) or spina bifida (SB).

DETAILED DESCRIPTION:
The overarching goal of this five-year, phase II, randomized clinical trial is to improve poor long-term health outcomes in both adolescents and young adults (AYA) with either a kidney transplant (KT) or spina bifida (SB), respectively. More specifically, this study will focus on decreasing premature allograft loss in subjects with kidney transplant (KT) due to medication nonadherence and kidney damage in subjects with SB due to urinary non-continence. To achieve these goals, this study will implement a real-time feedback system, Way to Health (WTH), that will provide education and support, increase awareness and incentivize positive health behavior, in addition to standard of care. Further, this study will investigate the mechanisms of behavior change by examining the role of financial incentives, positive feedback and the relationship between the two. The study will compare two cohorts of KT and SB subjects, which will undergo varied levels of financial incentives and positive feedback. Data from KT and SB subjects will be analyzed jointly and separately. This innovative mobile health (mhealth) strategy will improve our current measures of adherence and increase our understanding of factors that influence adherence for two AYA populations, KT and SB subjects, respectively. The study will contribute novel insight to inform the design of future interventions targeting persistence of behavior change and can be used in other centers and for other chronic disease groups.

The study intervention will use the WTH web-based platform to support AYA with KT or SB as they navigate their daily treatment burdens. This will be achieved via bi-directional text messaging, including the sending of reminders and positive feedback by WTH and the messaging of pictures of medication or catheter in hand at time of treatment by the participant. This intervention will assess sustainability of this novel bi-directional messaging system and the impact of providing education and support, increasing awareness and incentivizing positive health behavior in real-time.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 12-24 years.
2. Kidney Transplant subjects must be greater than 3 months post-transplant.
3. Spina Bifida subjects must be able to perform Clean Intermittent Catheterization (CIC) as part of their treatment.
4. Able to speak and read in English.
5. Willing and able to provide informed assent or consent.
6. Parental/guardian permission (informed consent) if appropriate.

Exclusion Criteria:

1. Unwilling to participate.
2. Unable to speak or read in English.
3. Unable to provide informed assent or consent.
4. Severe cognitive impairment, as reported by treating team in recruiting clinic.
5. On dialysis.
6. Acquired post-transplant lymphoproliferative disease less than one year prior to enrollment
7. Less than 3 months post-transplant.
8. Unable to perform CIC.
9. Prescribed Immunosuppressive medications once per day.
10. Provider recommendations of CIC once per day

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 465 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Amaral, MD, MHS, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (6):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data beyond those involved in the research study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from June 2017-April 2021. Potential participants were recruited from nephrology, urology, and Spina Bifida outpatient clinics either in person or over the phone.
Pre-assignment Details: After consenting to be a part of the study, participants were required to complete a set of baseline questionnaires before being assigned to a study arm. If a participant did not complete the questionnaires, they were not allowed to continue.
Groups:
- KT Arm 1 - No Feedback, Minimum Incentive: Subjects will receive daily text message reminders and report real-time treatment adherence with photos. They will receive compensation to encourage real-time adherence reporting. Subjects will also be able to log into a personal dashboard with a visual display of their weekly adherence performance and educational resources related to their primary disease. Every month, participants will receive a text encouraging them to visit their personal dashboard. The dashboard is able to track usage of the modules by individual. Parents/legal guardians will have access to these same educational materials via their own portals. Additionally, to mitigate the minimal risk of this study, parents/legal guardians will be notified if their child is excessively non-adherent.
  Behavioral Feedback and Economic Incentives: Arm 1: The purpose of this study is to determine the effectiveness of behavioral feedback plus economic incentives to promote treatment adherence among a large diverse population of adolescents and young adults (AYA) with kidney transplants (KT). In Arm 1, participants will not receive personalized feedback, nor will they receive the "extra" incentive of $10 for meeting their adherence goal.
- KT Arm 2 - Feedback, Maximum Incentive: Subjects will receive daily text message reminders and report real-time treatment adherence with photos, and will have web access to the educational modules through their portal. Every month, participants will receive a text encouraging them to visit their portals. In contrast to Arm 1, they will receive their weekly performance results by text to their phone with tailored feedback. In Arm 2, subjects will receive a larger incentive if they perform their desired treatment behavior. Incentive notification will be texted to participants. Similarly to Arm 1, parents/legal guardians will have access to the same educational materials via their own WTH portals. Additionally, to mitigate the minimal risk of this study, parents/legal guardians will be notified if their child is excessively non-adherent.
  Behavioral Feedback and Economic Incentives: Arm 2: The purpose of this study is to determine the effectiveness of behavioral feedback plus economic incentives to promote treatment adherence among a large diverse population of adolescents and young adults (AYA) with kidney transplants (KT). In Arm 2, participants will receive personalized feedback, and an "extra" incentive of $10 for meeting their adherence goal.
- SB Arm 1- No Feedback, Minimum Incentive: Subjects will receive daily text message reminders and report real-time treatment adherence with photos. They will receive compensation to encourage real-time adherence reporting. Subjects will also be able to log into a personal dashboard with a visual display of their weekly adherence performance and educational resources related to their primary disease. Every month, participants will receive a text encouraging them to visit their personal dashboard. The dashboard is able to track usage of the modules by individual. Parents/legal guardians will have access to these same educational materials via their own portals. Additionally, to mitigate the minimal risk of this study, parents/legal guardians will be notified if their child is excessively non-adherent.
  Behavioral Feedback and Economic Incentives: Arm 1: The purpose of this study is to determine the effectiveness of behavioral feedback plus economic incentives to promote treatment adherence among a large diverse population of adolescents and young adults (AYA) with spina bifida (SB). In Arm 1, participants will not receive personalized feedback, nor will they receive the "extra" incentive of $10 for meeting their adherence goal.
- SB Arm 2- Feedback, Maximum Incentive: Subjects will receive daily text message reminders and report real-time treatment adherence with photos, and will have web access to the educational modules through their portal. Every month, participants will receive a text encouraging them to visit their portals. In contrast to Arm 1, they will receive their weekly performance results by text to their phone with tailored feedback. In Arm 2, subjects will receive a larger incentive if they perform their desired treatment behavior. Incentive notification will be texted to participants. Similarly to Arm 1, parents/legal guardians will have access to the same educational materials via their own WTH portals. Additionally, to mitigate the minimal risk of this study, parents/legal guardians will be notified if their child is excessively non-adherent.
  Behavioral Feedback and Economic Incentives: Arm 2: The purpose of this study is to determine the effectiveness of behavioral feedback plus economic incentives to promote treatment adherence among a large diverse population of adolescents and young adults (AYA) with spina bifida (SB). In Arm 2, participants will receive personalized feedback, and an "extra" incentive of $10 for meeting their adherence goal.
Period: Intervention Phase
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive | SB Arm 1- No Feedback, Minimum Incentive | SB Arm 2- Feedback, Maximum Incentive
Started | 77 | 78 | 52 | 51
Completed | 67 | 73 | 49 | 44
Not Completed | 10 | 5 | 3 | 7
Not completed — Withdrawal by Subject | 7 | 2 | 3 | 7
Not completed — Developed exclusionary criteria | 3 | 3 | 0 | 0
Period: Follow-Up Phase
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive | SB Arm 1- No Feedback, Minimum Incentive | SB Arm 2- Feedback, Maximum Incentive
Started | 67 | 73 | 49 | 44
Completed | 66 | 68 | 45 | 39
Not Completed | 1 | 5 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 4 | 4 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Developed exclusionary criteria | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive | SB Arm 1- No Feedback, Minimum Incentive | SB Arm 2- Feedback, Maximum Incentive | Total
Number analyzed (Participants) | 77 | 78 | 52 | 51 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (2.9) | 16.8 (2.7) | 17.3 (2.9) | 16.7 (3.4) | 16.8 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 40 | 33 | 26 | 131
  Male | 45 | 38 | 19 | 25 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 7 | 5 | 31
  Not Hispanic or Latino | 66 | 70 | 45 | 46 | 227
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 2 | 3 | 6 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 14 | 8 | 6 | 44
  White | 46 | 57 | 28 | 38 | 169
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 11 | 4 | 9 | 4 | 28
Region of Enrollment [Number; unit: participants]
  United States | 77 | 78 | 52 | 51 | 258

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Subjects With Adherence Behavior Greater Than or Equal to 85% From Baseline and Intervention Period (6-month)
Description: Participants who do not submit the correct number of pictures within the prescribed window of their expected time due for treatment will be counted as non-adherent for that episode of med taking/cathing. The mean percentage of participants who achieved 85% adherence was calculated for each week from baseline (week 1) to the end of the 6 month time point (week 26).
Time Frame: baseline to 6 months
Population: These analyses followed the intention to treat principle.
Measure: Mean (Standard Deviation); unit: percentage of subjects
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive | SB Arm 1- No Feedback, Minimum Incentive | SB Arm 2- Feedback, Maximum Incentive
Number analyzed (Participants) | 77 | 78 | 52 | 51
percentage of subjects | 30.56 (0.08) | 42.04 (0.05) | 6.39 (0.03) | 12.14 (0.02)

2. Primary Outcome: Study Efficacy of Use of Way to Health Portal System
Description: Statistical analysis of the number and timing of messages sent to the Way to Health portal as well as how often the participants used the portal will determine study efficacy.
Time Frame: 12.5 months
Population: No data were collected on how often the participants used the portal. Only data on how often they utilized the text messaging portion of the program was collected and these were analyzed as part of adherence (primary outcome measure 1).
Arm/Group | Arm 1 - No Feedback, Minimum Incentive | Arm 2 - Feedback, Maximum Incentive
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Pressure Per Unit Volume of Bladder of Spina Bifida Subjects
Description: Urodynamic studies (UDS) in spina bifida subjects will test the change in bladder wall compliance, i.e. the change in pressure per unit volume of the bladder.
Time Frame: 12.5 months
Population: This secondary outcome could not be analyzed because urodynamic studies were very inconsistently performed on our subjects at each site. In order to calculate change in pressure per unit volume of the bladder, at least two urodynamic studies much be performed per patient. There were no patients who had two urodynamic studies performed so change could not be calculated and this outcome could not be analyzed.
Arm/Group | SB Arm 1- No Feedback, Minimum Incentive | SB Arm 2- Feedback, Maximum Incentive
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Coefficient of Variation (CV) of Immunosuppressive Drug Levels (Tacrolimus or Sirolimus) Between the Baseline (run-in) and Intervention Period.
Description: The difference between the coefficient of variation (CV) of immunosuppressive drug levels in kidney transplant patients at baseline and intervention period (6 months). CV was calculated using the average of three values of immunosuppressive drug levels at each time point. The change was calculated as the difference in mean value between baseline and 6 months.
Time Frame: baseline and at 6 months
Population: In order to calculate the coefficient of variation of immunosuppressive drug levels, three values are needed at each time point. Those that did not have three values at either time point could not be analyzed. Therefore the number of participants analyzed is less than the number randomized to each group.
Measure: Mean (Standard Deviation); unit: change in coefficient of variation
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive
Number analyzed (Participants) | 40 | 42
change in coefficient of variation | 4.69 (23.68) | 0.25 (23.19)

5. Other Pre Specified Outcome: Executive Function
Description: Behavior Rating Inventory of Executive Function questionnaire will be administered and answers will be analyzed.
Time Frame: 12.5 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Perceived Treatment Barriers - Spina Bifida
Description: The Spina Bifida and Cathing Barriers measure will be administered and answers will be analyzed.
Time Frame: 12.5 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mean Change in Perceived Adherence Behaviors as Measured by the Adolescent Medication Barriers Scale From Baseline to Intervention Period (6 Months)
Description: The Adolescent Medication Barrier Scale will be administered to the kidney transplant patients and answers will be analyzed. The Adolescent Medication Barriers Scale (AMBS) endorsement score is the sum of 17 items (rated 1,2,3=0, rated 4 & 5=1). The higher the endorsement score (range of 0-17) indicates that the adolescent perceived themselves as having more barriers to medication adherence.
Time Frame: Baseline to 6 months
Population: In order to calculate change between baseline and 6 months, KT participants needed to complete the AMBS measure at both timepoints. If the survey was missing at 6 months, they were not included in the analyses which is why the participants analyzed does not match the randomized number. This scale was only applicable to the KT cohort since we were measuring cathing adherence with the SB cohort and not medication adherence.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive
Number analyzed (Participants) | 45 | 45
score on a scale | 0.40 (2.32) | 0.27 (2.21)

8. Other Pre Specified Outcome: Change in Self-Efficacy Score From Baseline to Intervention Period (6 Month)
Description: Self-Efficacy for Managing Chronic Disease 6-Item Scale ranging from 1 (not at all confident) to 10 (totally confident). Total score is the mean of the 6-tems. The higher the score, the more self-efficacy. The outcome measure is the change in score 6 months-baseline.
Time Frame: baseline to 6 months
Population: In order to calculate change, the Self-efficacy for Managing Chronic Disease questionnaire needed to be answered at both the baseline and 6 month time points. If missing at either timepoint, they were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive | SB Arm 1- No Feedback, Minimum Incentive | SB Arm 2- Feedback, Maximum Incentive
Number analyzed (Participants) | 45 | 44 | 34 | 16
score on a scale | -0.38 (1.92) | 0.23 (2.12) | 0.1 (1.59) | -0.8 (1.77)

9. Other Pre Specified Outcome: Treatment Responsibility
Description: Allocation of Treatment Responsibility and the Sharing of Spina Bifida Management Responsibilities surveys will be administered and answers will be analyzed.
Time Frame: 12.5 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Disease Knowledge Score From Baseline to Intervention (6 Months)
Description: The Heart Transplant Knowledge questionnaire, adapted for Kidney Transplant patients, and the Knowledge of Spina Bifida survey will be administered and answers will be analyzed. There are 20 questions, each correct question = 1, each incorrect question =0. The total score ranges from 0-20. The higher the score, the more knowledge the participant has. The outcome measure will measure the change in score from 6 months to baseline.
Time Frame: baseline to 6 months
Population: The change in knowledge score can only be calculated if the participant completes the questionnaire at both the baseline and 6 month timepoints. If it is missing at either timepoint, they were not included in the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KT Arm 1 - No Feedback, Minimum Incentive | KT Arm 2 - Feedback, Maximum Incentive | SB Arm 1- No Feedback, Minimum Incentive | SB Arm 2- Feedback, Maximum Incentive
Number analyzed (Participants) | 45 | 45 | 39 | 29
score on a scale | -0.29 (2.71) | 0 (2.79) | 0.92 (4.84) | 1.1 (5.14)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the duration of a subject's participation in the study, which was one year.
Description: There is no greater than minimal risk to subjects in this study. Any AE associated with the study protocol would be immediately reported to the DSMB, the PIs and the IRB. If the AE was not considered related to the study protocol, it did not need to be reported. We confirm there were no participant deaths that occurred during the course of the study. All SAEs and AEs reported here were collected as hospitalizations that occurred during the study and none were considered related to the study.
Arm/Group | Arm 1 - No Feedback, Minimum Incentive | Arm 2 - Feedback, Maximum Incentive
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/129
Serious Adverse Events (participants affected / at risk) | 32/129 | 34/129
Other Adverse Events (participants affected / at risk) | 32/129 | 38/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - No Feedback, Minimum Incentive (N=129) | Arm 2 - Feedback, Maximum Incentive (N=129)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 3 (3)
Bowel Dysfunction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Headaches (General disorders) | 0 (0) | 2 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (2)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 3 (4) | 2 (2)
Other Renal Related (Renal and urinary disorders) | 3 (4) | 5 (7)
Pain (General disorders) | 1 (1) | 1 (3)
Paraesophageal Hiatal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 3 (8) | 0 (0)
Scoliosis (Nervous system disorders) | 0 (0) | 1 (1)
Shunt issue (Nervous system disorders) | 2 (3) | 4 (4)
Spinal (Nervous system disorders) | 1 (1) | 2 (2)
Surgery (Surgical and medical procedures) | 4 (4) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0)
Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Issue (Renal and urinary disorders) | 3 (4) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - No Feedback, Minimum Incentive (N=129) | Arm 2 - Feedback, Maximum Incentive (N=129)
Acute Illness (General disorders) | 13 (16) | 12 (14) — Can include fever, abdominal pain, vomitting, diarrhea)
Concern for rejection (Renal and urinary disorders) | 12 (21) | 14 (26) — Can include acute rejection, elevated creatinine, IVIG infusion
Urinary Tract Infection Related (Renal and urinary disorders) | 7 (12) | 12 (14)

LIMITATIONS AND CAVEATS:
Due to issues with recruitment, our final sample size is likely underpowered. Low response rates for some of our study surveys also prevented us from having enough data to analyze some of our secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03045276/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03045276/ICF_001.pdf